CLINICAL TRIAL: NCT00662649
Title: An Extension of the 24-month, Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Comparing Efficacy and Safety of Fingolimod (FTY720) 1.25 mg and 0.5 mg Administered Orally Once Daily Versus Placebo in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Long-term Efficacy and Safety of Fingolimod (FTY720) in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2301E1; 2007-004122-24 (EudraCT Number)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis.; Relapse-remitting; Fingolimod
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Fingolimod 1.25 mg (Experimental): Patients continued the same dose to which they had been randomized in the Core study (CFTY720D2301/NCT00289978), fingolimod 1.25 mg/day, in this Extension study.
  Interventions: Drug: Fingolimod 1.25 mg
- Fingolimod 0.5 mg (Experimental): Patients continued the same dose to which they had been randomized in the Core study, fingolimod 0.5 mg/day, in this Extension study.
  Interventions: Drug: Fingolimod 0.5 mg
- Placebo-fingolimod (Experimental): Patients randomized to placebo in the Core study were re randomized to fingolimod (either 0.5 or 1.25 mg/day) in this Extension study.
  Interventions: Drug: Fingolimod 0.5 mg; Drug: Fingolimod 1.25 mg
- Placebo-fingolimod 1.25 mg (Experimental): Patients randomized to placebo in the Core study were re randomized to fingolimod 1.25 mg/day in this Extension study.
  Interventions: Drug: Fingolimod 1.25 mg
- Placebo-fingolimod 0.5 mg (Experimental): Patients randomized to placebo in the Core study were re randomized to fingolimod 0.5 mg/day in this Extension study.
  Interventions: Drug: Fingolimod 0.5 mg

INTERVENTIONS:
Drug: Fingolimod 0.5 mg — Patients self-administered fingolimod 0.5 mg capsules orally once daily.
  Other Names: FTY720
  Arms: Fingolimod 0.5 mg; Placebo-fingolimod; Placebo-fingolimod 0.5 mg
Drug: Fingolimod 1.25 mg — Patients self-administered fingolimod 1.25 mg capsules orally once daily.
  Other Names: FTY720
  Arms: Fingolimod 1.25 mg; Placebo-fingolimod; Placebo-fingolimod 1.25 mg

SUMMARY:
This extension study of was designed to evaluate the long-term safety, tolerability, and efficacy of fingolimod (FTY720) in patients with multiple sclerosis. The Extension study was an extension to the 24-month Core study (CFTY720D2301/NCT00289978).

ELIGIBILITY:
Inclusion Criteria:

* Patients should complete the 24 month core study

Exclusion Criteria:

* Patients with other chronic disease of the immune system, malignancies, acute pulmonary disease, cardiac failure, etc.
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 920 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (103):
- Australia (5):
  - Novartis Investigative Site, Chatswood
  - Novartis Investigative Site, Fitzroy
  - Austin Health, Department of Neurology, Heidelberg
  - Novartis Investigative Site, North Gosford
  - Novartis Investigative Site, Woodville
- Belgium (7):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Overpelt
  - Novartis Investigative Site, Sijsele - Damme
  - Novartis Investigative Site, Sint-Truiden
- Canada (8):
  - Novartis Investigative Site, Halifax
  - Novartis Investigative Site, Kingston
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Nepean
  - Novartis Investigative Site, Regina
  - Novartis Investigative Site, Toronto
  - Novartis Investigative Site, Vancouver
- Czechia (8):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Plzen - Lochotin
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Rychnov nad Kněžnou
  - Novartis Investigative Site, Teplice
- Novartis Investigative Site, Talinn, Estonia
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (9):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Athens, Greece
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Székesfehérvár
- Novartis Investigative Site, Dublin, Ireland
- Israel (4):
  - Novaratis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Safed
- Netherlands (6):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard
  - Novartis Investigative Site, Tilburg
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Romania (4):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Lasi
  - Novartis Investigative Site, Tg. Mures
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (3):
  - Novartis Investigational Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigational Site, Žilina
- South Africa (3):
  - Novartis Investigational Site, Cape Town
  - Novartis Investigational Site, Rosebank
  - Novartis Investigational Site, Umhlanga
- Sweden (2):
  - Novartis Investigational Site, Gothenburg
  - Novartis Investigational Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (8):
  - Novartis Investigational Site, Ankara
  - Novartis Investigational Site, Bursa
  - Novartis Investigational Site, Cerrahpasa/Istanbul
  - Novartis Investigational Site, Gaziantep
  - Novartis Investigational Site, Istanbul
  - Novartis Investigational Site, Izmir
  - Novartis Investigational Site, Mersin
  - Novartis Investigational Site, Yenisehir/Izmir
- United Kingdom (5):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sheffield

REFERENCES:
- See also: Fingolimod clinical trials information website — http://www.msclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1272 patients randomly assigned to treatment in the Core study (ClinicalTrials.gov ID NCT00289978), 1033 completed the 24-month double-blind treatment phase and were eligible to enter the Extension study. A total of 920 of the 1033 patients entered the Extension study and received treatment.
Groups:
- Fingolimod 1.25 mg: Patients continued the same dose to which they had been randomized in the core study, fingolimod 1.25 mg/day, in this extension study.
- Placebo: Patients randomized to placebo in the Core study who were subsequently re-randomized to fingolimod(either 1.25 or 0.5 mg/day) in the Extension study.
- Placebo-fingolimod 0.5: Patients randomized to placebo in the core study were re randomized to fingolimod 0.5 mg/day in this extension study.
Period: Core Study (24 Months)
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5
Started | 429 | 425 | 418 | 0 (This reporting group is used only in extension study.) | 0 (This reporting group is used only in extension study.)
Intent to Treat (ITT) | 429 | 425 | 418 | 0 | 0
Completed | 332 | 369 | 332 | 0 | 0
Not Completed | 97 | 56 | 86 | 0 | 0
Not completed — Withdrawal by Subject | 31 | 17 | 28 | 0 | 0
Not completed — Adverse Event | 22 | 13 | 18 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 13 | 6 | 25 | 0 | 0
Not completed — Abnormal laboratory value(s) | 20 | 9 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 5 | 7 | 0 | 0
Not completed — Protocol Violation | 5 | 5 | 4 | 0 | 0
Not completed — Abnormal test procedure result(s) | 2 | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 2 | 0 | 0
Period: Extension Study (Month 24 to 60)
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5
Started | 289 | 331 | 0 (This reporting group is used only for core study) | 145 | 155
Extension Intent to Treat Population | 287 | 330 | 0 | 145 | 154
From Beginning of Core at Month 24 | 289 | 331 | 0 | 145 | 155
From Beginning of Core at Month 30 | 276 | 324 | 0 | 136 | 152
From Beginning of Core at Month 36 | 270 | 311 | 0 | 130 | 145
From Beginning of Core at Month 42 | 254 | 301 | 0 | 120 | 136
From Beginning of Core at Month 48 | 125 | 152 | 0 | 58 | 67
From Beginning of Core at Month 54 | 31 | 32 | 0 | 11 | 13
Completed | 245 ("completed" refers to patients that completed extension study in different time points.) | 290 | 0 | 112 | 126
Not Completed | 44 | 41 | 0 | 33 | 29
Not completed — Abnormal laboratory value(s) | 10 | 5 | 0 | 8 | 3
Not completed — Abnormal test procedure result(s) | 3 | 1 | 0 | 1 | 3
Not completed — Administrative problems | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 6 | 9 | 0 | 6 | 10
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Subject withdrew consent | 19 | 23 | 0 | 15 | 9
Not completed — Subject no longer requires study drug | 0 | 1 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 3 | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg | Total
Number analyzed (Participants) | 289 | 331 | 145 | 155 | 920
Age Continuous [Mean (Standard Deviation); unit: years] — All demographic measurements are based on extension randomized/safety population.
  years | 37.2 (8.87) | 36.5 (8.60) | 36.6 (9.21) | 38.1 (8.26) | 37.0 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 234 | 107 | 106 | 651
  Male | 85 | 97 | 38 | 49 | 269

OUTCOME MEASURES:

1. Primary Outcome: Annualized Aggregate Relapse Rate (ARR) During Months 0 to End of Study(Core [CFTY720D2301/NCT00289978] and Extension Study)
Description: ARR is defined as the number of confirmed relapses in a year. A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection. The annualized ARR for each treatment group was the mean of the annualized ARRs for all patients in the group, calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25.
Time Frame: Months 0 to end of study (maximum up to 60 months)
Population: Core Intent to treat (ITT) population: All patients who were randomized in the Core study and received at least 1 dose of Core study drug.
Measure: Number (95% Confidence Interval); unit: Relapses per year
Groups:
- Placebo-fingolimod: Patients randomized to placebo in the Core study who were subsequently re-randomized to FTY720 (either 1.25 or 0.5 mg/day) in the Extension study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod
Number analyzed (Participants) | 429 | 425 | 418
Relapses per year | 0.164 [0.138 to 0.195] | 0.185 [0.158 to 0.217] | 0.357 [0.310 to 0.411]

2. Secondary Outcome: Change in Mean Number of New or Newly Enlarged T2 Magnetic Resonance Imaging (MRI) Lesions During Months 0-24 (Core Study) and Months 24-48 (Extension Study)
Description: The number of new or newly enlarged T2 lesions was assessed with T2-weighted MRI scans. A T2-weighted MRI scan utilizes particular values of the echo time (TE) and the repetition time (TR) parameters of image acquisition. Inflammation and tissue damage are seen as bright areas in T2 images and are often referred to as T2 lesions. T2 weighted MRI scans are a sensitive way to evaluate the brain for demyelinating diseases, such as multiple sclerosis.
Time Frame: Months 0-24 (core study) and Months 24-48 (extension study)
Population: Extension intent-to-treat (ITT) population: All extension randomized patients that received at least 1 dose of extension study drug. The analysis included number of patients with evaluable T2 MRI scans.
Measure: Mean (Standard Deviation); unit: Lesions
Groups:
- Placebo-fingolimod 1.25 mg: Patients randomized to placebo in the core study were re-randomized to fingolimod 1.25 mg/day in this extension study.
- Placebo-fingolimod 0.5 mg: Patients randomized to placebo in the core study were re-randomized to fingolimod 0.5 mg/day in this extension study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Number analyzed (Participants) | 123 | 163 | 64 | 69
Lesions
  Months 0-24 | 2.14 (5.234) | 2.66 (9.395) | 12.83 (17.573) | 8.12 (11.083)
  Months 24-48 | 1.71 (4.902) | 2.58 (9.256) | 2.34 (4.745) | 1.43 (2.446)
  Change from Months 0-24 to Months 24-48 | -0.43 (4.393) | -0.09 (7.423) | -10.48 (15.980) | -6.68 (9.876)

3. Primary Outcome: Time to First Confirmed Relapse up to End of Study: Kaplan-Meier Estimate of Percentage of Patients Relapse-free
Description: A relapse was confirmed when it was accompanied by an increase of at least half a step (0.5) on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS). Kaplan-Meier estimates of the percentage of relapse-free patients at end of study and and 95% confidence intervals (CIs) were presented for the treatment groups.
Time Frame: Core baseline to end of study (maximum up to 60 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod
Number analyzed (Participants) | 429 | 425 | 418
Percentage of patients | 59.85 [53.90 to 65.80] | 59.29 [54.17 to 64.41] | 37.18 [32.15 to 42.22]

4. Secondary Outcome: Percentage of Patients Free of New or Newly Enlarged T2 Magnetic Resonance Imaging (MRI) Lesions During Months 0-24 (Core Study) and Months 24-48 (Extension Study)
Description: as for outcome 2
Time Frame: Months 0-24 (core study) and Months 24-48 (extension study)
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Number analyzed (Participants) | 126 | 163 | 65 | 69
Percentage of patients
  Months 0-24 | 53.2 | 50.3 | 18.5 | 23.2
  Months 24-48 | 57.1 | 69.3 | 52.3 | 55.1

5. Secondary Outcome: Percent Change in Brain Volume From Month 0 to Month 24 (Core Study) and From Month 24 to Month 48 (Extension Study)
Description: Calculations of brain volume change were performed using the structural image evaluation of normalized atrophy (SIENA), software included in the Functional Magnetic Resonance Imaging of the Brain (FMRIB) software library. SIENA is a fully automated method for estimating temporal brain volume change.
Time Frame: Months 0-24 (core study) and Months 24-48 (extension study)
Population: Extension intent-to-treat (ITT) population: All extension randomized patients that received at least 1 dose of extension study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Number analyzed (Participants) | 287 | 330 | 145 | 154
Percent change
  Month 0 to Month 24, n=75, 109, 41, 49 | -1.011 (1.3477) | -0.983 (1.6291) | -1.511 (1.6401) | -1.419 (1.3923)
  Month 24 to Month 48, n=75, 109, 41, 49 | -0.871 (1.4164) | -0.780 (1.9266) | -1.103 (1.4073) | -0.903 (1.1406)

6. Primary Outcome: Annualized Aggregate Relapse Rate (ARR) During Months 0-24 (Core Study) and Months 24-48 (Extension Study)
Description: as for outcome 1
Time Frame: Months 0-24 (core study) and Months 24-48 (extension study)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Relapses per year
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Number analyzed (Participants) | 287 | 330 | 145 | 154
Relapses per year
  Months 0-24 | 0.064 [0.043 to 0.094] | 0.111 [0.084 to 0.148] | 0.301 [0.230 to 0.393] | 0.292 [0.222 to 0.383]
  Months 24-48 | 0.074 [0.051 to 0.108] | 0.095 [0.070 to 0.128] | 0.164 [0.117 to 0.231] | 0.130 [0.092 to 0.184]

7. Primary Outcome: Change (Expressed as Ratio) in the Annualized Aggregate Relapse Rate (ARR) From Months 0-24 (Core Study) to Months 24-48 (Extension Study)
Description: as for outcome 1
Time Frame: Months 0-24 (core study) and Months 24-48 (extension study)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Ratio of relapses per year
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Number analyzed (Participants) | 287 | 330 | 145 | 154
Ratio of relapses per year | 1.164 [0.830 to 1.633] | 0.850 [0.658 to 1.099] | 0.547 [0.390 to 0.767] | 0.446 [0.320 to 0.620]

8. Secondary Outcome: Percent Change in Brain Volume From Month 0 End of Study (Core and Extension Study)
Description: as for outcome 5
Time Frame: Months 0 to end of study (maximum up to 60 months)
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core study and received at least 1 dose of Core study drug. This analysis included only patients with value at both core baseline and end of study.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Placebo-fingolimod: Patients randomized to placebo in the Core study who were subsequently re-randomized to fingolimod (either 1.25 or 0.5 mg/day) in the Extension study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod
Number analyzed (Participants) | 250 | 299 | 259
Percent change | -1.639 (1.9265) | -1.674 (2.1182) | -2.241 (2.1873)

9. Secondary Outcome: Time to First 3-month Confirmed Disability Progression up to End of Study Based on Expanded Disability Status Scale (EDSS): Kaplan-Meier Estimate of Percentage of Patients Free of Disability Progression
Description: Kurtzke's Expanded Disability Status Scale (EDSS) is a scale for assessing neurologic impairment in multiple sclerosis (MS) includes a series of scores in each of eight functional systems such as Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, Cerebral, and Other. The EDSS steps range from 0 (normal) to 10 (death due to MS). The Kaplan-Meier estimates of the percentage of participants free of disability progression at end of study and their 95% CIs were provided for each treatment group.
Time Frame: Core baseline to end of study (maximum up to 60 months)
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core study and received at least 1 dose of Core study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Placebo-fingolimod: Patients randomized to placebo in the Core study who were subsequently re-randomized to fingolimod(either 1.25 or 0.5 mg/day) in the Extension study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod
Number analyzed (Participants) | 429 | 425 | 418
Percentage of patients | 74.15 [69.54 to 78.75] | 73.90 [69.44 to 78.37] | 66.28 [61.28 to 71.28]

ADVERSE EVENTS:
Description: Safety reported on extension safety population which includes all patients who received at least 1 dose of Extension study drug. Patients were analyzed according to the actual treatment received during extension.
Groups:
- Fingolimod 1.25mg: Patients randomized to fingolimod 1.25 mg/day in the Core study. These patients continued the same dose in the Extension study.
- Fingolimod 0.5mg: Patients randomized to fingolimod 0.5 mg/day in the Core study. These patients continued the same dose in the Extension study.
- Placebo-Fingolimod 1.25mg: Patients randomized to placebo in the Core study who were subsequently re-randomized to fingolimod 1.25 mg/day in the Extension study.
- Placebo-Fingolimod 0.5mg: Patients randomized to placebo in the Core study who were subsequently re-randomized to fingolimod 0.5 mg/day in the Extension study.
Arm/Group | Fingolimod 1.25mg | Fingolimod 0.5mg | Placebo-Fingolimod 1.25mg | Placebo-Fingolimod 0.5mg
Serious Adverse Events (participants affected / at risk) | 31/289 | 31/331 | 17/145 | 11/155
Other Adverse Events (participants affected / at risk) | 236/289 | 273/331 | 107/145 | 130/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25mg (N=289) | Fingolimod 0.5mg (N=331) | Placebo-Fingolimod 1.25mg (N=145) | Placebo-Fingolimod 0.5mg (N=155)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Genital infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Crush injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 3 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 | 0
Personality disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lymphomatoid papulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Selective abortion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Vascular stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25mg (N=289) | Fingolimod 0.5mg (N=331) | Placebo-Fingolimod 1.25mg (N=145) | Placebo-Fingolimod 0.5mg (N=155)
Lymphopenia (Blood and lymphatic system disorders) | 52 | 52 | 18 | 17
Diarrhoea (Gastrointestinal disorders) | 14 | 29 | 10 | 10
Fatigue (General disorders) | 12 | 23 | 7 | 8
Bronchitis (Infections and infestations) | 19 | 20 | 10 | 11
Cystitis (Infections and infestations) | 7 | 12 | 8 | 3
Gastroenteritis (Infections and infestations) | 15 | 11 | 3 | 5
Influenza (Infections and infestations) | 30 | 33 | 9 | 12
Nasopharyngitis (Infections and infestations) | 82 | 84 | 39 | 44
Oral herpes (Infections and infestations) | 19 | 24 | 10 | 11
Pharyngitis (Infections and infestations) | 14 | 17 | 8 | 5
Sinusitis (Infections and infestations) | 8 | 15 | 7 | 10
Upper respiratory tract infection (Infections and infestations) | 39 | 58 | 23 | 24
Urinary tract infection (Infections and infestations) | 20 | 27 | 12 | 8
Alanine aminotransferase increased (Investigations) | 10 | 11 | 16 | 9
Carbon monoxide diffusing capacity decreased (Investigations) | 21 | 16 | 10 | 9
Gamma-glutamyltransferase increased (Investigations) | 7 | 8 | 12 | 8
Lymphocyte count decreased (Investigations) | 29 | 16 | 12 | 14
Weight decreased (Investigations) | 3 | 6 | 4 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 18 | 24 | 7 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 21 | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 21 | 12 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 18 | 9 | 8
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 16 | 4 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 10 | 5 | 3
Dizziness (Nervous system disorders) | 7 | 7 | 6 | 10
Headache (Nervous system disorders) | 27 | 41 | 18 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 13 | 11
Hypertension (Vascular disorders) | 24 | 18 | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.